CLINICAL TRIAL: NCT00814645
Title: A Placebo-Controlled, Phase 1b, Dose-Finding, Safety, Pharmacodynamic Effect Study of Sodium Nitrite Inhalation Solution (AIR001 INHALATION SOLUTION) in Normal, Healthy Volunteers
Brief Title: Dose-Finding, Safety, Pharmacodynamic Effect Study of Sodium Nitrite Inhalation Solution in Normal, Healthy Volunteers
Acronym: AIR001-CS02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aires Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIR001 CS02
Record Dates: First submitted 2008-12-22; First posted 2008-12-25 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose level 1 (Active Comparator): a single dose (5 mg sodium nitrite)of AIR001 Inhalation Solution administered by inhalation following nebulization
  Interventions: Drug: Sodium Nitrite Inhalation Solution
- Dose level 2 (Active Comparator): a single dose(15 mg sodium nitrite) of AIR001 Inhalation Solution administered by inhalation following nebulization
  Interventions: Drug: Sodium Nitrite Inhalation Solution
- Dose level 3 (Active Comparator): a single dose(45 mg sodium nitrite) of AIR001 Inhalation Solution administered by inhalation following nebulization
  Interventions: Drug: Sodium Nitrite Inhalation Solution
- Dose level 4 (Active Comparator): a single dose(113 mg sodium nitrite) of AIR001 Inhalation Solution administered by inhalation following nebulization
  Interventions: Drug: Sodium Nitrite Inhalation Solution
- Expansion arm (Placebo Comparator): On Day 1, subjects will receive a single placebo-form dose of inhaled nebulized AIR001 Inhalation Solution (containing diluent and excipient solutions alone). On Day 2, the same subjects will receive a single administration of AIR001 Inhalation Solution at the minimum pharmacologically active and safe dose identified from dose levels 1-4. Subjects will be blinded to the treatment schema.
  Interventions: Drug: Placebo and AIR001 Inhalation Solution (Expansion arm)

INTERVENTIONS:
Drug: Sodium Nitrite Inhalation Solution — a single dose of AIR001 Inhalation Solution administered by inhalation following nebulization
  Other Names: AIR001 Inhalation Solution
  Arms: Dose level 1; Dose level 2; Dose level 3; Dose level 4
Drug: Placebo and AIR001 Inhalation Solution (Expansion arm) — On Day 1, subjects will receive a single placebo-form dose of inhaled nebulized AIR001 Inhalation Solution (containing diluent and excipient solutions alone). On Day 2, the same subjects will receive a single administration of AIR001 Inhalation Solution at the minimum pharmacologically active and safe dose identified from dose levels 1-4. Subjects will be blinded to the treatment schema.
  Other Names: AIR001 Inhalation Solution
  Arms: Expansion arm

SUMMARY:
This study is designed to investigate the safety and tolerability of AIR001 Inhalation Solution when administered under conditions of hypoxia and to identify dose levels of drug resulting in a reduction in pulmonary arterial pressure under these hypoxic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Normal male and female volunteers
* Age 18-55
* Demonstrate a rise in pulmonary artery pressure to low inspired oxygen concentration (a normal response to breathing a low level of oxygen)

Exclusion Criteria:

* Significant medical illnesses
* Risk factors for pulmonary hypertension
* G6PD or Cytochrome B5 Reductase deficiencies
* History of any form of altitude sickness
* Current prescription or over the counter medication use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The measurement of pulmonary arterial pressures by echocardiography. | Pretreatment and up to 2 hours post treatment

SECONDARY OUTCOMES:
Plasma pharmacokinetics | Pretreatment to 8 hours post treatment
Hematology, blood chemistry, coagulation and urinalysis, methemoglobin, oxygen saturation, electrocardiogram, troponin, and vital signs and adverse events. | Pretreatment, post treatment, and 24 hours post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne K Swan, M.D., Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States